CLINICAL TRIAL: NCT03982316
Title: Telehealth Behavioral Migraine Management
Acronym: TeleBMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10345; UL1TR002556 (NIH)
Record Dates: First submitted 2019-06-08; First posted 2019-06-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Behavioral Migraine Management (Experimental): Participants will receive weekly online education sessions in the following categories: Relaxation, Early Warning Signs, Triggers, Medication Adherence, Reducing Migraine Impact, Stress Management, Biofeedback, and Relapse Prevention. Participants will receive four monthly 50-minute telehealth sessions with a doctoral psychology student in a clinical health psychology program covering these topics, and three check-ins to enhance adherence to behavior change strategies. Participants will complete a daily headache diary throughout the course of treatment.
  Interventions: Behavioral: Telehealth Behavioral Migraine Management

INTERVENTIONS:
Behavioral: Telehealth Behavioral Migraine Management — 1) Weekly online modules; 2) Monthly 50 minute telephone calls; 3) 3 15-minute telephone check ins.

SUMMARY:
This project aims to develop the protocol and obtain feasibility and acceptability information for Telehealth Behavioral MIgraine Management in a single-arm pre-post pilot study. The investigator and study team aim to recruit 20 people with migraine from the Montefiore Headache Center in the Bronx NY. Participants will receive the 12-week protocol including a mobile app headache diary, an online patient manual with interactive vignettes, 4 50-minute telehealth sessions, and 3 15-minute check-ins.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of migraine
* Current self-reported symptoms meeting the International Classification for Headache Disorders -- 3 criteria for migraine
* Self-reported between 4 and 20 headache days/month
* Aged 18-65
* Can read English
* Capacity to consent

Exclusion Criteria:

* Psychiatric illness that would interfere with study participation
* Meeting criteria for probable medication overuse headache

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of TeleBMM | Week 0 through Week 12
  Number of treatment components participants complete (out of 20)

SECONDARY OUTCOMES:
Patient-rated satisfaction | Post-treatment survey at Week 12
  Patient-rated satisfaction (acceptability) with the program on a Likert-type scale ranging from 0 ("Not at all satisfied") to 4 ("Very satisfied")
Quality of Life (Migraine Specific) | Change from Pre-treatment (Week 0) to Post-treatment (Week 12)
  Score on the MSQ v 2.1, a 14-item survey assessing quality of life in people with migraine.
Headache frequency | Slope change from Week 0 to Week 12
  Participants complete a daily headache diary, on which each 7 day week they denote whether they have had a headache attack.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Seng, Ph.D., Principal Investigator — Yeshiva University/Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No